CLINICAL TRIAL: NCT01870336
Title: Combination of Lateral Foot Orthoses and Knee Brace for Treatment of the Medial Knee Osteoarthritis
Brief Title: Combination of Lateral Foot Orthoses and Knee Brace for Treatment of the Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Fonds de la Recherche en Santé du Québec (Other Government); Ergorecherche Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OC-2013
Record Dates: First submitted 2013-05-23; First posted 2013-06-06 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lateral customized foot orthoses (Experimental): Foot orthoses with arch support and lateral inclination set at 7° (alone)
  Interventions: Device: Combined treatment of medial knee osteoarthritis
- Knee brace (Experimental): OdrA Knee brace (alone)
  Interventions: Device: Combined treatment of medial knee osteoarthritis
- Combination of the two treatments (Experimental): Combination of Lateral customized foot orthoses and knee brace
  Interventions: Device: Combined treatment of medial knee osteoarthritis

INTERVENTIONS:
Device: Combined treatment of medial knee osteoarthritis

SUMMARY:
The purpose of this study is to evaluate the immediate and short-term effects of the combination of lateral customized foot orthoses on the pain and medial knee loading during gait among medial knee osteoarthritis patients. The effects of the combination is compared to the single use of these devices. The investigators recruited 22 knee osteoarthritis. They have to wear each of treatments (foot orthoses, knee brace and combination) during three months. A fifteen days wash-out period is given after each three months. Biomechanical evaluation is carried out before and after each three months. This evaluation consisted of three questionnaires (Knee Osteoarthritis Outcome Score (KOOS), Western Ontario and McMaster Universities Osteoarthritis Index ( WOMAC) and Medical Outcome Study Short Form-36( MOS-SF36)), a motion analysis with an optoelectronic system, then a 6-min walk test. During motion analysis, ten gait trials are executed without treatment and ten with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic medial knee OA (Kellgren-Lawrence grade I, II or III) according to clinical and radiological criteria of the American College of Rheumatology
* Knee pain > 31/100 (Western Ontario and McMaster Universities Arthritis Index - WOMAC)
* Moderately active
* Varus knee alignment equal or superior to 2°

Exclusion Criteria:

* Severe knee OA (K-L grade IV)
* Rheumatoid arthritis or other inflammatory arthritis
* Avascular necrosis
* History of periarticular fracture or septic arthritis
* Bone metabolic disease
* Pigmented villonodular synovitis
* Cartilaginous disease
* Neuropathic arthropathy
* Synovial osteochondromatosis
* Total or partial knee arthroplasty
* Flexion contracture of ipsi- or contra-lateral knee greater than 15°
* Hip or ankle joint damage with mobility limitation
* Obesity (BMI ≥ 40)
* Intra-articular corticosteroids injection in the affected knee during the two previous months
* Reduced mobility (Charnley class C)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Knee adduction moment | Change from Baseline at 3 months
Change in Knee pain | Change from Baseline at 3 months
  A 20-cm visual analog scale (0-100) is used to assess pain.

SECONDARY OUTCOMES:
Change in Spatiotemporal gait parameters | Change from Baseline at 3 months
Change in Knee adduction angle | Change from Baseline at 3 months
Change in Comfort | Change from Baseline at 3 months
  A 20-cm visual analog scale (0-100) is used to assess comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Corbeil, PhD, Study Director — Laval University; Yoann Dessery, MSc, Principal Investigator — Laval University; Étienne L Belzile, MD, Study Director — Laval University
Locations (1):
- Pavillon de l'Éducation Physique et des Sports - Université Laval, Québec, Quebec, Canada